CLINICAL TRIAL: NCT02742038
Title: Effectiveness of Fluoride Varnish in the Prevention of Early Childhood Caries in Non-fluoridated Areas: A 24-month Randomized Controlled Trial
Brief Title: Effectiveness of Fluoride Varnish in the Prevention of Early Childhood Caries: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Patricia Muñoz Millán, Staff, Universidad de La Frontera
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FON11-0002; SA1154 (Other: CONICYT)
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoride varnish plus education (Experimental): Biannual fluoride varnish every 6 month/ 24 months plus educational component
  Interventions: Other: Fluoride varnish plus education
- Placebo varnish plus education (Placebo Comparator): Biannual placebo varnish every 6 month/ 24 months plus educational component
  Interventions: Other: Fluoride varnish plus education

INTERVENTIONS:
Other: Fluoride varnish plus education — Biannual varnish every 6 month/ 24 months plus educational component

SUMMARY:
Triple-blind randomized controlled trial with two parallel arms conducted between 2012 and 2014. Children 2-3 years old, from 28 rural public preschools, located in low socioeconomic areas of Chile were invited to participate. Oral health education component was given to children, parents and educators, twice yearly. A new toothbrush and toothpaste for each child was delivered to the parents at baseline and in each of the follow-up visits. The experimental group was treated with fluoride varnish every six months while the control group received placebo applications. 277 preschoolers (2 to 3 years) Main outcome: Number of Caries Incident Cases, increment dmft index

DETAILED DESCRIPTION:
Triple-blind randomized controlled trial with two parallel arms conducted between 2012 and 2014. Children 2-3 years old, from 28 rural public preschools, located in low socioeconomic areas of Chile were invited to participate. Oral health education component was given to children, parents and educators, twice yearly. A new toothbrush and toothpaste for each child was delivered to the parents at baseline and in each of the follow-up visits. The experimental group was treated with fluoride varnish every six months while the control group received placebo applications. A trained, calibrated dentists blinded to treatment arm performed a visual-tactile dental assessment at 6, 12, 18 and 24 months. The number of incidents children with caries were recollected as the number of caries during the follow-up visits.

Nº of participant/ centres: 277 preschoolers (2 to 3 years) of 28 public preschools in non-fluoridated areas.

Main outcome: Number of Caries Incident Cases, increment dmft index

ELIGIBILITY:
Inclusion Criteria:

* Children between 24 an 47 months, free of caries, preschooler of a public centre and living in a non-fluoridated community.

Exclusion Criteria:

* Children compromised medically, or with developmental or learning disabilities, or with a temporary residence or with dental developmental anomalies.

Ages: 24 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 275 (Actual)
Dates: Start 2012-03; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Dental Caries | 24 months
  Number of caries and incident cases

SECONDARY OUTCOMES:
Caries increment | 24 months
  caries increment measured by the amount of change in dmfs index from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Zaror, Master, Study Director — Universidad de La Frontera; María José Martínez, Doctor, Study Chair — Cochrane; Patricia Muñoz, Master, Study Chair — U. Frontera

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Munoz-Millan P, Zaror C, Espinoza-Espinoza G, Vergara-Gonzalez C, Munoz S, Atala-Acevedo C, Martinez-Zapata MJ. Effectiveness of fluoride varnish in preventing early childhood caries in rural areas without access to fluoridated drinking water: A randomized control trial. Community Dent Oral Epidemiol. 2018 Feb;46(1):63-69. doi: 10.1111/cdoe.12330. Epub 2017 Aug 29. PMID 28850712